CLINICAL TRIAL: NCT02127307
Title: An Open-Label, Multicenter, Phase 4 Study to Demonstrate the Prognostic Usefulness of AdreView™ Scintigraphy for Identifying Subjects With Heart Failure Who Will Experience Death During 60 Months Follow-up.
Brief Title: Phase 4 Study to Demonstrate Prognostic Usefulness of AdreView™ Scintigraphy for Identifying Subjects With Heart Failure Who Will Experience Death During 60 Months Follow-up.
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: H2O Clinical LLC (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-122-016
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure (HF)
Keywords: Myocardial sympathetic innervation; Heart failure (HF); Nuclear imaging; Radiopharmaceutical
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This aim of the study is to investigate the prognostic usefulness of AdreView™ imaging to identify those subjects with New York Heart Association (NYHA) Class II or III HF who will die during 60 months of follow-up from the date of administration of AdreView™ in prior studies MBG311, MBG312, or MBG312C (hereafter included in MBG312).

ELIGIBILITY:
Inclusion Criteria:

* The subject was a HF subject who had signed informed consent for MBG311 or MBG312.
* The subject was administered AdreView™ in MBG311 or MBG312.
* The subject completed the late planar imaging assessments (at a minimum) required by the protocols for MBG311 and MBG312, and those images were read and judged diagnostic by at least 2 blinded readers.
* In addition, all subjects must meet 1 of the following 3 inclusion criteria.
* If the subject can be located, he/she provides informed consent to allow the investigator access to medical records and/or gives permission for the investigator to speak to treating physicians.
* If the subject can be located and he/she declines to provide informed consent, the IRB/EC provides a waiver of consent to allow the investigator to record that the subject is alive.
* If the subject cannot be located, the IRB/EC provides a waiver of consent to allow the investigator to access available medical records for care provided subsequent to last date of subject participation in MBG311, MBG312, and/or MBG313 and/or to allow collection of data from publicly available sources.

Exclusion Criteria:

* The subject withdrew or was withdrawn from MBG311 or MBG312 because of a protocol violation.
* The subject underwent heart transplantation during MBG311, MBG312, or MBG313.
* The subject was recorded to have died during MBG311, MBG312, or MBG313.
* The subject voluntarily withdrew from MBG311, MBG312, or MBG313, and the IRB/EC has not provided a waiver to allow recording of subject survival status in such an instance.
* The subject cannot be located, cannot be contacted, and no information can be found to establish survival status beyond the date of last contact in MBG311, MBG312, or MBG313, including information available as a result of an IRB/EC-approved waiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients (NYHA Class II or III) with left ventricular ejection fraction ≤35% at time of enrolment in MBG311 or MBG312.
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Zubeldia, M.D., Study Chair — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the present study GE-122-016 (NCT02127307), participants previously administered AdreView™ (123ImIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) were followed to identify who died during 60 months of follow-up from the date of administration of 123I-mIBG.
Pre-assignment Details: Of 964 heart failure (HF) participants included in the efficacy population of MBG311 (NCT00126425) and MBG312 (NCT00126438), 694 were contacted in this study as 101 participants died and 169 were not contacted due to participant consent not obtained and/or some sites declined to participate.
Groups:
- AdreView™- Heart Failure Group: HF participants who were administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) were observed to identify who died during 60 months of follow-up at 6-month intervals from the date of administration of 123I-mIBG.
Period: Overall Study
Arm/Group | AdreView™- Heart Failure Group
Started | 964
Completed | 656
Not Completed | 308
Not completed — Protocol Violation | 36
Not completed — Lost to Follow-up | 2
Not completed — Death | 101
Not completed — Other than specified above | 169

BASELINE CHARACTERISTICS:
Arm/Group | AdreView™- Heart Failure Group
Number analyzed (Participants) | 964
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 772

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between the Occurrence of Death and 123I-mIBG Uptake on Planar Scintigraphy With Heart to Mediastinum (H/M) Ratio of <1.60 vs H/M ≥1.60
Description: H/M ratio for 123I-mIBG uptake at 3 hours 50 minutes post administration was calculated by dividing the counts/pixel in the total myocardium region of interest (ROI) by the counts/pixel in the 7x7 pixel mediastinal ROI. H/M ratios were categorized as 'Low' and 'High' based on being <1.6 or ≥1.6 respectively. The efficacy of 123I-mIBG was based on the prognostic value of the imaging data, as reflected by the H/M ratio, for identifying HF participants at lower risk of death during 60 months of follow-up.
Time Frame: From the date of administration of 123I-mIBG in studies MBG-311 or MBG-312 up to 60 months
Population: Efficacy population was 961 participants who received investigational medicinal product (IMP) and had a diagnostic 3 hour 50 minute planar image in MBG311 or MBG312. Here, 'n' signifies number of participants with available data for specified category.
Measure: Number; unit: number of death or other adverse events
Arm/Group | AdreView™- Heart Failure Group
Number analyzed (Participants) | 961
number of death or other adverse events
  Participants with H/M ratio <1.60 (n=760) | 292
  Participants with H/M ratio ≥1.60 (n=201) | 42
Statistical Analysis 1: Comparison: AdreView™- Heart Failure Group; AdreView-Heart Failure Group with H/M <1.60 vs. H/M ≥1.60: Data analysis was performed using Cox proportional hazards model to demonstrate the relationship of consensus numeric H/M ratio and time to adverse cardiac events to identify participants with higher risk of death. Hazard (risk) of a death for a participant with H/M ratio at time "t" was expressed as Hl (t)/Hh (t)=Ψ,where Hl (t) and Hh (t) denote the hazard of an event at time t for participants with low H/M and high H/M respectively; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — At 0.025 level of significance; Hazard Ratio (HR) = 0.4460, 95% CI 2-sided [0.3227 to 0.6156]

ADVERSE EVENTS:
Time Frame: From the date of administration of 123I-mIBG in studies MBG-311 or MBG-312 up to 60 months
Description: The main objective of the study was to monitor participants previously administered AdreView™ (123ImIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) to identify participants who died up to 60 months from the date of administration of 123I-mIBG, therefore, no safety evaluations performed in this study
Arm/Group | AdreView™- Heart Failure Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.